CLINICAL TRIAL: NCT04221594
Title: Quantification of Myocardial Blood Flow Using Dynamic PET/CTA Fused Imagery to Determine the Physiological Significance of Specific Coronary Lesions.
Brief Title: Quantification of Myocardial Blood Flow Using Dynamic PET/CTA Fused Imagery
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Samsung Medical Center (Other); Seoul National University (Other); Chonnam National University Hospital (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Marina Piccinelli, Principal Investigator, Emory University
Other Study IDs: IRB00107151; 1R01HL143350-01 (NIH)
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Coronary Artery Disease
Keywords: Fractional flow reserve; Myocardial blood flow; Relative flow reserve; Non-invasive measure; Cardiac catheterization; CT coronary angiography; Dynamic PET; Invasive coronary angiography; 3D fusion dPET/CTA; FFRCT
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CAD detection/risk assessment: Patients with angina referred for the assessment of CAD will undergo imaging studies to develop tools to fuse coronary anatomic data obtained from CCTA with dPET data to non-invasively measure absolute MBF, MFR and RFR along vessels centerlines and across coronary lesions.
  Interventions: Procedure: Invasive Cardiac Catheterization (ICA); Procedure: Coronary Computed Tomographic Angiogram (CCTA); Procedure: Dynamic Cardiac Positron Emission Tomography (dPET)

INTERVENTIONS:
Procedure: Invasive Cardiac Catheterization (ICA) — Invasive functional measurements will be performed to assess the functional significance of specific lesions by means of FFR and CFR, and to test the presence of microvascular disease by means of IMR in all vessels for which the procedures are feasible. In summary, a 5- to 7-F guide catheter without side holes is used to engage the coronary artery and a pressure-temperature sensor-tipped guidewire introduced. The pressure sensor is positioned at the distal segment of a target vessel, and intracoronary nitroglycerine (100-200 mg) administered before each measurement. The best systolic and diastolic phase (located between 30-50%, and 60-75% of the cardiac cycle) will be selected for successive processing as it allows a relative motion free visualization of the main vessels and the myocardium.
Procedure: Coronary Computed Tomographic Angiogram (CCTA) — Fasting patients will undergo a test for coronary calcium by CT; calcium scoring analysis will be done post image data acquisition using the manufacturer's software. Nitroglycerine will be administered in all patients (sublingual administration prior to CCTA initiation). CT acquisitions will be prospectively ECG-gated (30-80% of the cardiac cycle). The acquisition begins with a scout scan to identify the borders of the heart to minimize the field of view and exposure to the patient. A bolus of 60 mL nonionic contrast agent is then injected followed by 60 mL of saline at a rate of 4 mL/s to enhance signal from coronary arteries and blood chambers. In case of irregular heart rate, beta-blockers can be provided to keep optimal heart rate ~65-70 bpm. Trans-axial images are reconstructed by means of a filtered back-projection algorithm.
Procedure: Dynamic Cardiac Positron Emission Tomography (dPET) — Patients will be asked to fast for 24 hours prior to the test. Before the resting perfusion phase, a single low-dose CT-based transmission scan is acquired for attenuation correction (AC) of all subsequent acquisitions. AC-CT images are automatically registered to the perfusion images, visually verified and manually corrected if necessary. Resting perfusion imaging started with the intravenous injection of a single bolus of 82Rb. Pharmacological stress imaging is obtained after adenosine infusion (140 μg/kg/min) through a peripheral vein, followed by a second dose of 82Rb. Image reconstruction is achieved by means of ordered subset expectation maximization (OSEM) iterative method. The hemodynamic responses to rest/stress tests are collected in terms of mean heart rate, mean blood systolic pressures and diastolic at rest and stress. Dynamic, gated and ungated trans-axial reconstructions are saved in DICOM format for further analysis and processing.

SUMMARY:
This observational prospective clinical study is to develop software tools to fuse coronary anatomy data obtained from CT coronary angiography with dynamic PET data to noninvasively measure absolute myocardial blood flow, flow reserve and relative flow reserve across specific coronary lesions. Results will be compared to those obtained invasively in the catheterization laboratory.

DETAILED DESCRIPTION:
This observational prospective clinical study is to develop software tools to fuse coronary anatomy data obtained from CT coronary angiography with dynamic PET data to noninvasively measure absolute myocardial blood flow, flow reserve and relative flow reserve across specific coronary lesions. These results will be compared to those obtained invasively in the catheterization laboratory. The long-term objective of the study is to improve the care of cardiac patients by developing, validating and implementing clinically computer-based methods to noninvasively determine the physiological significance of specific coronary lesions using methods to fuse and quantify multi-modality cardiac imagery.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years of age) - as the research topic to be studied is irrelevant to children
* Written consent form
* Patients with prior dynamic PET or CCTA or ICA for any indications

Exclusion Criteria:

* Previous history of allergy to iodinated contrast
* Previous CABG
* Serum creatinine levels >1.8 mg/dl unless patient has end stage kidney disease, not producing any urine and dialysis
* History of claustrophobia (CT tunnel length of more than 100 cm)
* Significant arrhythmias or tachycardia
* History of frequent asthma attacks or acting wheezing
* Second- and third-degree heart block
* Systolic blood pressure of < 90 mmHg
* Heart failure with NYHA class III-IV at the time of the CCTA procedure. If it is deemed that, the heart failure has been resolved or the patient was incorrectly labeled as having heart failure the radiology physician in charge will verify the absence of Heart Failure at the time of CCTA and perform the procedure.
* Recent myocardial infarction
* If the patient has been diagnosed with unstable angina within 24 hours prior to CCTA, the patient will not be consented. If the patient does not have the diagnosis of unstable angina and is consented, the radiology physician in charge will verify the absence of unstable angina at the time of CCTA.
* Patients enrolled and consented for the invasive measurements that at the time of catheterization exhibit severe vessel disease and/or obstructions that prevent the operator from safely conducting the measurements will be removed from the study; further research imaging sessions - if planned - will be canceled and patients indicated as "screen failure" in our enrollment log.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with angina referred to an initial imaging test for the assessment of CAD will be screened and considered for inclusion in the study. Different hospital policies and guidelines determine which initial test is commonly requested: at Emory University Hospital patients who underwent a dPET will be considered for enrollment; at the South Korean centers patients who received a CTA will be screened. Depending on test results, patients who are referred to undergo a cardiac catheterization, will be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Myocardial blood flow (MBF) measurement comparing non-invasive to the traditional approaches | Up to 3 months
  Myocardial blood flow (MBF) measured in milliliters per minute per gram of tissue is providing unique pathophysiologic and diagnostic information on the function of the coronary macro- and microcirculation.
Vessel-specific quantification of myocardial blood flow RFR | Up to 3 months
  Ratio of absolute hyperemic MBFs (abnormal / normal) measured in mL/min/g.

SECONDARY OUTCOMES:
Absolute myocardial blood flow (MBF) measurement comparing non-invasive to the traditional approaches | Up to 3 months
  Absolute myocardial blood flow (MBF) measured in ml/min/gm provides incremental diagnostic and prognostic information over relative perfusion alone.
Myocardial flow reserve (MFR) measurement comparing non-invasive to the traditional approaches | Up to 3 months
  Myocardial flow reserve (MFR) provide incremental diagnostic and prognostic information over relative perfusion alone.
Fractional Flow Reserve (FFR) measurement comparing non-invasive to the traditional approaches | Up to 3 months
  FFR calculates the maximum flow down a vessel in the presence of stenosis compared to maximum flow in the hypothetical absence of the stenosis.
Stress myocardial blood flow (sMBF)/Regional myocardial blood flow (rMBF) ratio | Up to 3 months
  Stress myocardial blood flow (sMBF)/Regional myocardial blood flow (rMBF) ratio will be calculated
Distal/proximal pressure ratio | Up to 3 months
  Distal/proximal pressure ratio will be calculated
Discriminatory power of dPET/CTA. And FFR(CTA) | Up to 3 months
  Predictive discriminatory power of each technique will be compared to ICA (FFR)

CONTACTS AND LOCATIONS:
Overall Officials: Marina Piccinelli, PhD, Principal Investigator — Emory University
Locations (6):
- United States (3):
  - Emory Clinic, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Saint Francis Hospital & Heart Center, Roslyn, New York
- South Korea (3):
  - Chonnam National University, Gwangju
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
All PET imaging data, All CTA imaging data, Invasive Coronary Angiography (ICA) static images used for measurements, all processing and measurements made from all imaging data, patient pertinent demographics and clinical data, as well as dictionary of database formats will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Processed anonymized data and extracted measurements are available now to co-investigators as each evaluable case is completed. All raw data described above is also available to co-investigators now on demand and will be accessible to the co-investigators remotely as soon as the imaging database is operational expected to be online, password protected on May 1, 2020. The same data described in the above paragraph will be available to all others (non-co-investigators) two years after termination of this grant cycle, August 1, 2024.
Access Criteria: All data is available to all co-investigators now and all others on 8/1/2024.Co-investigators will analyze and test the hypotheses listed in the R01 proposal. Priority for testing the scientific/technical hypotheses will be given to the Emory investigators and those for testing the clinical hypotheses to the external investigators. Other project sub-analysis will be prioritized on a first come first served basis when approved by each of the grant site principal investigators. All others can analyze the data for any purpose starting on 8/1/2024. All shared anonymized data will be available from password protected imaging databases and databases of extracted measurements and clinical demographics databases via a Gmail/Gdrive account being constructed.

REFERENCES:
- [Derived] AlBadri A, Piccinelli M, Cho SG, Lee JM, Jaber W, De Cecco CN, Samady H, Koo BK, Bom HS, Garcia EV. Rationale and design of the quantification of myocardial blood flow using dynamic PET/CTA-fused imagery (DEMYSTIFY) to determine physiological significance of specific coronary lesions. J Nucl Cardiol. 2020 Jun;27(3):1030-1039. doi: 10.1007/s12350-020-02052-0. Epub 2020 Feb 5. PMID 32026327

DOCUMENTS (1):
  • Informed Consent Form (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT04221594/ICF_000.pdf